CLINICAL TRIAL: NCT07226414
Title: Evaluating the Impact of Perelel Prenatal on Biomarkers in Healthy Pregnant Women.
Brief Title: Prenatal Study in Healthy Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Perelel Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AFCRO-200
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy
MeSH Terms: interventions — Prenatal Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal Capsules (Experimental): Prenatal serving is 2 capsules + one omega softgel
  Interventions: Dietary Supplement: Prenatal Capsule
- Gummy Prenatal (Active Comparator): Prenatal serving is 2 gummies that also contains omega
  Interventions: Dietary Supplement: Prenatal Gummy

INTERVENTIONS:
Dietary Supplement: Prenatal Capsule — This study will look at the impacts of a prenatal capsule vs a gummy comparator prenatal. The prenatal consists of 2 multivitamin + micronutrient blend with one omega softgel.
  Other Names: Perelel Prenatal
  Arms: Prenatal Capsules
Dietary Supplement: Prenatal Gummy — This prenatal gummy is a commercially available multivitamin that also contains omega-3 DHA and EPA
  Arms: Gummy Prenatal

SUMMARY:
Clinical Trial Summary

The goal of this clinical trial is to address the impact of a gummy prenatal vs a capsule based prenatal in pregnant women. The main question it aims to answer is:

Does 12-week daily administration of Prenatal Capsule affect serum iron levels in pregnant women in their second trimester compared to a comparator gummy prenatal?

Researchers will compare Prenatal Capsule to a comparator Prenatal Gummy to see if there are differences in serum iron levels after 12 weeks of daily use.

Participants will:

Take their assigned prenatal supplement (either Prenatal Capsule or the comparator Prenatal Gummy) daily for 12 weeks Be in their second trimester of pregnancy during the study period Have their serum iron levels measured at baseline and after the 12-week intervention period

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent.
* Healthy pregnant women between 21- 40 years of age (inclusive).
* Pregnant women in the second trimester of pregnancy (gestational age of 14-19 weeks).
* Willing to consume the Study Product daily for the duration of the study.

Exclusion Criteria:

* History of drug or alcohol abuse
* Is hypersensitive to any of the contents of the study product, that would preclude intake of the study products.
* Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk, or would confound the interpretation of the study results as judged by the investigator on the basis of medical history.
* Severe nausea and vomiting in the first trimester, including hyperemesis gravidarum (HG)
* Inability to tolerate oral supplement intake due to gastrointestinal symptoms during the first trimester of pregnancy
* Prior Pregnancy Complications (gestational diabetes (GD), HG, or pre-eclampsia, NTDs (Neural Tube Defects))
* Current pregnancy complications (GD, Iron Deficiency Anemia)
* Hypertension
* Diabetes mellitus
* Cardiovascular disease
* Class II/III obesity (defined as BMI ≥35.0 Kg/m2)
* Malabsorption syndromes (e.g., celiac disease, inflammatory bowel disease)
* Severe anemia or iron overload disorders
* Thyroid disorders
* Current or recent (in the past 12 weeks prior to Visit 1) use of a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results, as judged by the investigator. Prohibited medications include:

Medications that contain fat-soluble vitamins A, E, or K in high doses

- Current or recent (in the past 12 weeks prior to Visit 1) use of prohibited nutritional or non-nutritional supplements that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results as judged by the investigator.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Requires biological females (pregnancy)
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to end of intervention on iron levels | 12 weeks
  Serum iron will be measured as primary outcome

SECONDARY OUTCOMES:
Change from baseline to end of intervention on folate status | 12 weeks
  Change from baseline (Day 1) to end of intervention in Prenatal capsule compared to Comparator product on red blood cell folate
Change from baseline to end of intervention on omega-3 status | 12 weeks
  Change from baseline (Day 1) to end of intervention (Day 85) in Prenatal capsule compared to Comparator product on:
  Red Blood Cell (RBC) Omega-3 Index (% Total Omega-3 Fatty Acids) Docosahexaenoic acid (DHA) as a percentage of RBC omega-3 fatty acids Eicosapentaenoic acid (EPA) as a percentage of RBC omega-3 fatty acids
Change from baseline to end of intervention on serum Vitamin D | 12 weeks
  Change from baseline (Day 1) to end of intervention (week 12) in Prenatal capsule compared to Comparator product on Serum Vitamin D (25-hydroxyvitamin D (25(OH)D)
Change from baseline to end of intervention on choline status | 12 weeks
  Change from baseline (Day 1) to end of intervention (Day 85) in Prenatal capsule compared to Comparator product on: Plasma choline, Plasma betaine, and Plasma zinc

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Clinical Trials, Chicago, Chicago, Illinois, United States